CLINICAL TRIAL: NCT06977620
Title: Effect of Closed Kinetic Chain and Weight Shifting Exercises on Postural Stability in Unilateral Post Mastectomy Lymphedema
Brief Title: Effect of CKC and WS Exercises on Postural Stability in Unilateral Post Mastectomy Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Kamal Mousa Mohamed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005746
Record Dates: First submitted 2025-05-03; First posted 2025-05-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Postmastectomy Lymphedema
Keywords: postural stability; closed kinetic chain exercises; weight shifting exercises
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: The study will be four-armed, single-blind (participant), parallel-group, randomized control trial. Sixty patients who have unilateral post mastectomy lymphedema will participate in this study. Their ages will range from 40 to 60 years. The patients will be subdivided randomly into four equal groups by using simple randomization technique 1:1 ratio to four equal groups according to sample size calculation
Who Masked: Participant
Masking Description: single-blind (participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (CKC group) (Active Comparator): This group will include 15 patients who will receive closed kinetic chain exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. CDT includes (skin care, manual lymphatic drainage, compression bandages, compression garments and exercises). The total exercise time will be 30 minutes, three times per week for eight weeks.
  Interventions: Other: Closed kinetic chain exercises; Other: Complete Decongestive Therapy
- Group B (WS group): (Active Comparator): This group will include 15 patients who will receive weight shifting exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. The total exercise time will be 30 minutes, three times per week for eight weeks.
  Interventions: Other: Weight shifting exercises; Other: Complete Decongestive Therapy
- Group C (Combined group) (Active Comparator): This group will include 15 patients who will receive closed kinetic chain and Weight shifting exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. The total exercise time will be 60 minutes; 30 minutes of CKC and 30 minutes of WS exercise three times per week for eight weeks
  Interventions: Other: Closed kinetic chain exercises; Other: Weight shifting exercises; Other: Complete Decongestive Therapy
- Group D (control group) (Placebo Comparator): This group will include 15 patients who will receive complex decongestive therapy (CDT) for the treatment of lymphedema. CDT includes (skin care, manual lymphatic drainage, compression bandages, compression garments and exercises).
  Interventions: Other: Complete Decongestive Therapy

INTERVENTIONS:
Other: Closed kinetic chain exercises — Closed kinetic chain (CKC) exercises emphasize weight-bearing movements where the distal segment of the extremity is fixed, and motion occurs as the proximal segment moves over the stabilized distal segment.
  Other Names: CKC
  Arms: Group A (CKC group); Group C (Combined group)
Other: Weight shifting exercises — Weight-shifting is a crucial aspect of dynamic postural control, which refers to the ability to maintain one's bodyweight within the base of support. Lateral weight-shifting, in particular, is essential for maintaining posture under dynamic conditions and is commonly performed in various activities of daily living
  Other Names: WS
  Arms: Group B (WS group):; Group C (Combined group)
Other: Complete Decongestive Therapy — CDT includes (skin care, manual lymphatic drainage, compression bandages, compression garments and exercises).
  Other Names: CDT

SUMMARY:
Post-mastectomy lymphedema is one of the most common chronic complications that significantly impacts patients' quality of life following breast cancer surgery. postural stability is maintained through the intricate integration of muscular forces, sensory input from mechanoreceptors, and biomechanical feedback. closed kinetic chain (CKC) exercises play a crucial role in enhancing musculoskeletal stability by countering gravitational forces during both rest and movement. weight shifting and balance are fundamental components of functional movement. Proprioceptive training, which focuses on improving body awareness and balance, is essential for developing trunk control

DETAILED DESCRIPTION:
Sixty patients who have unilateral post mastectomy lymphedema will participate in this study. Their ages will range from 40 to 60 years. The patients will be subdivided randomly into four equal groups.

1.1.a- Group A (n= 15) (CKC group): This group will include 15 patients who will receive closed kinetic chain exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. CDT includes (skin care, manual lymphatic drainage, compression bandages, compression garments and exercises). The total exercise time will be 30 minutes, three times per week for eight weeks.

1.1.b- Group B (n= 15) (WS group): This group will include 15 patients who will receive weight shifting exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. The total exercise time will be 30 minutes, three times per week for eight weeks.

1.1.c- Group C (n= 15) (Combined group): This group will include 15 patients who will receive closed kinetic chain and Weight shifting exercises, in addition to complex decongestive therapy (CDT) for the treatment of lymphedema. The total exercise time will be 60 minutes; 30 minutes of CKC and 30 minutes of WS exercise three times per week for eight weeks.

1.1.d- Group D (n= 15) (control group): This group will include 15 patients who will receive complex decongestive therapy (CDT) for the treatment of lymphedema. CDT includes (skin care, manual lymphatic drainage, compression bandages, compression garments and exercises).

ELIGIBILITY:
Inclusion Criteria:

Women who had a history of BCRS with upper limb lymphedema. • Age range of 40-60 years.

• The body mass index (BMI) is less than 30 Kg/m2.

• Consciousness and ability to communicate orally or in writing.

• Treatment by unilateral mastectomy with lymph node dissection.

• No obvious abnormal spine morphology or postural abnormalities visible to the naked eye.

• All participants had moderate lymphedema according to the lymphedema severity assessment.

Exclusion Criteria:

Patients with metastases. • Differences between lower limb length.

• Having acute or chronic vestibular, neurological, and orthopedic diseases.

• Surgery related to spine causing limitation of motion.

• Women with psychiatric disorders, reconstructive surgery.

• Bilateral mastectomy. Diagnosis with a neurological, skeletal, or rheumatic disorder or other disease that seriously affects body posture.

• History of bodily injury such as a spinal, shoulder, or neck injury, resulting in permanent alteration of the normal body posture prior to the unilateral mastectomy.

• Failure to complete follow-up for any reason over the course of the study.

• Peripheral polyneuropathy, cognitive dysfunction.

• Patients taking medication that affects body balance.

• Severe arthritis or orthopedic conditions in their lower extremity

• Poor conditioning, acute pain in any reason,

• Neurological disorders including visual problems.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who had a history of BCRS with upper limb lymphedema
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Kinesis Balance™ fall prevention app | Eight weeks
  Patients will be instructed to hold the phone firmly against their sternum and stand with their eyes open, in a semi-tandem stance, for 30 s. The app contains audio and visual instructions on how to prepare for and complete the test as well as an audio cue to indicate test start and stop.

SECONDARY OUTCOMES:
Time Up and Go Test (TUG) | Eight weeks
  Patients will be asked to stand up from a chair with armrests, walk three meters, turn, walk back, and sit down. The time taken to complete this task will be measured in seconds using a stopwatch
Functional Reach Test (FRT) | Eight weeks
  The patient will enter a standing position on a line marked on the floor. An inch tape will be attached to a wall at approximately shoulder height of the subject. The therapist will stand 5-10 feet away from the patient and instruct them to stand close to the wall without touching it, while facing the inch tape, with the shoulder flexed at 90° and the hand in a fist. The therapist will record the starting position at the knuckle of the third metacarpal head on the ruler. The patient will then be instructed to reach as far forward as possible along the length of the tape without moving their feet. The therapist will once again record the location of the knuckle of the third metacarpal.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamal, PHD, Principal Investigator — Teaching Assistant of Physical Therapy for Surgery Cairo University Egypt
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Publication at international journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January, 2027
Access Criteria: Open access

DOCUMENTS (1):
  • Study Protocol (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT06977620/Prot_000.pdf